CLINICAL TRIAL: NCT01493193
Title: Effects of Different Endurance Training Protocols on Physical Performance in Cardiac Patients
Brief Title: Different Endurance Training Protocols in Cardiac Rehabilitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Primar, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UISM-5
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Endurance Training; High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endurance training with constant work load (Active Comparator)
  Interventions: Other: Endurance training with constant work load
- Pyramid-Training (Experimental)
  Interventions: Other: Pyramid-Training
- High-intensity interval training (Experimental)
  Interventions: Other: High-intensity interval training

INTERVENTIONS:
Other: Endurance training with constant work load — Endurance training with constant work load(n=15): 31min at 65-75% HRmax
  Arms: Endurance training with constant work load
Other: Pyramid-Training — Pyramid-Training (n=15): One Pyramid consists of 8 one-minute blocks. Those are grouped starting with one block of 70-75% HRmax, followed by one block at 75-80% HRmax and another one at 80-85% HRmax. The top of the pyramid are 2 blocks of 85-90% HRmax. Intensity is lowered afterwards with one block at 80-85% HRmax, followed by one block at 75-80% HRmax and last one at 70-75% HRmax. Two more pyramids follow, each divided by 2min of active recovery at 65-70% HRmax, making it a total of 28min.
  Arms: Pyramid-Training
Other: High-intensity interval training — HIT (n=15): 4x4min intervals at 85-95% HRmax divided by 3x3min of active recovery at 60-70% HRmax, making it a total of 25min
  Arms: High-intensity interval training

SUMMARY:
It is the aim of the study to compare the effects of 6 weeks of either high-intensity interval training (HIT; carried out at correctly assessed 85-95% of maximal heart rate), pyramid, or continuous endurance training, on changes of physical exercise capacity in cardiac patients.

The three exercise arms (isocaloric) are composed as follows:

Endurance training (n=15): 31min at 65-75% HRmax; HIT (n=15): 4x4min intervals at 85-95% HRmax divided by 3x3min of active recovery at 60-70% HRmax, making it a total of 25min; Pyramids (n=15): One Pyramid consists of 8 one-minute blocks. Those are grouped starting with one block of 70-75% HRmax, followed by one block at 75-80% HRmax and another one at 80-85% HRmax. The top of the pyramid are 2 blocks of 85-90% HRmax. Intensity is lowered afterwards with one block at 80-85% HRmax, followed by one block at 75-80% HRmax and last one at 70-75% HRmax. Two more pyramids follow, each divided by 2min of active recovery at 65-70% HRmax, making it a total of 28min.

All protocols are initiated by 5min of warm-up and end with 5min of cool-down, both at 60-70% HRpeak.

Primary Outcome: Individual maximum power output in watt (Pmax). Secondary Outcome: Change of power output in watt at lactate thresholds at 2 and 4 mmol/l.

ELIGIBILITY:
Inclusion Criteria:

At least one of the following diagnoses within the previous 3 months:

* acute coronary syndrome (STEMI)
* acute coronary syndrome (NSTEMI)
* aortocoronary bypass surgery
* PCI
* stable coronary heart disease

Exclusion Criteria:

* Unstable angina pectoris
* Heart failure (NYHA IV)
* Acute endomyocarditis or other acute infections
* Pulmonary artery embolism or phlebothrombosis within the previous 6 months
* Hemodynamically unstable arrhythmia
* Hypertrophic cardiomyopathy
* participation in another study within the previous 6 months
* Medical conditions which prevent patients from complying with the exercise program

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Individual maximum power output in watt (Pmax) | 6 weeks
  Change of individual maximum power output in watt (Pmax) on a bicycle ergometer after the training intervention of controlled physical activity within 6 weeks

SECONDARY OUTCOMES:
Power output in watt at lactate threshold of 2 and 4 mmol/l | 6 weeks
  Change of power output in watt at lactate thresholds at 2 and 4 mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Josef Niebauer, MD, PhD, MBA, Study Chair — Paracelsus Medical University; Marcus Tschentscher, MSc, Principal Investigator — Paracelsus Medical University
Locations (1):
- Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University, Salzburg, Salzburg, Austria

REFERENCES:
- [Background] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Background] Niebauer J, Hambrecht R, Velich T, Hauer K, Marburger C, Kalberer B, Weiss C, von Hodenberg E, Schlierf G, Schuler G, Zimmermann R, Kubler W. Attenuated progression of coronary artery disease after 6 years of multifactorial risk intervention: role of physical exercise. Circulation. 1997 Oct 21;96(8):2534-41. doi: 10.1161/01.cir.96.8.2534. PMID 9355890
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Helgerud J, Hoydal K, Wang E, Karlsen T, Berg P, Bjerkaas M, Simonsen T, Helgesen C, Hjorth N, Bach R, Hoff J. Aerobic high-intensity intervals improve VO2max more than moderate training. Med Sci Sports Exerc. 2007 Apr;39(4):665-71. doi: 10.1249/mss.0b013e3180304570. PMID 17414804
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- See also: Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University Salzburg, Austria — http://www.salk.at/sportmedizin.html
- See also: Salzburg Regional Hospital — http://www.salk.at